CLINICAL TRIAL: NCT00942500
Title: Effects of Postconditioning On Myocardial Reperfusion in Patients With ST-segment Elevation Myocardial Infarction
Brief Title: Effects of Postconditioning On Myocardial Reperfusion
Acronym: POST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-02-007
Record Dates: First submitted 2009-07-13; First posted 2009-07-21 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Myocardial Reperfusion; Myocardial Infarction
Keywords: Post-conditioning; ST-elevation myocardial infarction; Angioplasty, Transluminal, Percutaneous Coronary
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Ischemic Postconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post-conditioning (Experimental)
  Interventions: Procedure: Post-conditioning
- Conventional primary PCI (No Intervention)

INTERVENTIONS:
Procedure: Post-conditioning — Coronary angiogram is performed to allow identification of the culprit coronary artery and to check no reperfusion before PCI (TIMI grade <2). Restoration of coronary blood flow can be achieved by thrombus aspiration, balloon angioplasty, direct stenting or together.In the postconditioning group, immediately after restoration (TIMI grade ≥2) of coronary flow (without regard to method of achieving restoration), angioplasty balloon will be positioned at the culprit lesion or stented segment and inflated 4 times for 1 minute with low-pressure (4 to 6 atm) inflations, each separated by 1 minute of reflow. When restoration of coronary flow is achieved by thrombus aspiration or balloon angioplasty and residual stenosis is remained ≥30%, stent will be deployed.
  Arms: Post-conditioning

SUMMARY:
The purpose of this study is to investigate the effects of postconditioning on myocardial reperfusion in patients with ST-segment elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria General Inclusion Criteria

* Subject must be at least 18 years of age.
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving postconditioning and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure
* Diagnosis of STEMI

  1. presence of chest pain for more than 30 minutes but less than 12 hours after symptom onset
  2. ST-segment elevation more than 1 mm in at least 2 contiguous leads

Angiographic Inclusion Criteria

* Target lesion(s) must be located in a native coronary artery
* Target lesion(s) must be amenable for percutaneous coronary intervention
* TIMI flow grade of infarct related arteries <2

General Exclusion Criteria

* Patients with hemodynamic instability or those with cardiogenic shock
* Target lesion is located in left main stem
* Rescue PCI after thrombolysis or facilitated PCI
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The dichotomous rate of complete ST-segment resolution (STR) | at 30 minutes after final contrast injection

SECONDARY OUTCOMES:
Myocardial blush grade | within 10 minutes after PCI
Thrombolysis in Myocardial Infarction (TIMI) flow grade | within 10 minutes after PCI
Angiographic no-reflow | during PCI
All death | at 30 days and 1 year
Stent thrombosis | at 30 days and 1 year
Cardiac death | at 30 days and 1 year
Myocardial infarction | at 30 days and 1 year
Severe heart failure | at 30 days and 1 year
  Severe heart failure was defined as heart failure with documented arterial partial pressure of oxygen less than 60 mmHg or with pulmonary edema documented radiographically or requiring intubation, 100% oxygen, or insertion of a mechanical support device.
Target vessel revascularization (TVR) | at 30 days and 1 year
Composite of death, MI, severe heart failure, or stent thrombosis | at 30 days and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hahn JY, Yu CW, Park HS, Song YB, Kim EK, Lee HJ, Bae JW, Chung WY, Choi SH, Choi JH, Bae JH, An KJ, Park JS, Oh JH, Kim SW, Hwang JY, Ryu JK, Lim DS, Gwon HC. Long-term effects of ischemic postconditioning on clinical outcomes: 1-year follow-up of the POST randomized trial. Am Heart J. 2015 May;169(5):639-46. doi: 10.1016/j.ahj.2015.01.015. Epub 2015 Feb 27. PMID 25965711
- [Derived] Kim EK, Hahn JY, Song YB, Lee SC, Choi JH, Choi SH, Lee SH, Choe YH, Gwon HC. Effect of ischemic postconditioning on myocardial salvage in patients undergoing primary percutaneous coronary intervention for ST-segment elevation myocardial infarction: cardiac magnetic resonance substudy of the POST randomized trial. Int J Cardiovasc Imaging. 2015 Mar;31(3):629-37. doi: 10.1007/s10554-015-0589-y. Epub 2015 Jan 15. PMID 25589306
- [Derived] Hahn JY, Song YB, Kim EK, Yu CW, Bae JW, Chung WY, Choi SH, Choi JH, Bae JH, An KJ, Park JS, Oh JH, Kim SW, Hwang JY, Ryu JK, Park HS, Lim DS, Gwon HC. Ischemic postconditioning during primary percutaneous coronary intervention: the effects of postconditioning on myocardial reperfusion in patients with ST-segment elevation myocardial infarction (POST) randomized trial. Circulation. 2013 Oct 22;128(17):1889-96. doi: 10.1161/CIRCULATIONAHA.113.001690. Epub 2013 Sep 25. PMID 24068776